CLINICAL TRIAL: NCT05435690
Title: Evaluation of a New Navigation System in Computer-assisted Total Knee Arthroplasty
Acronym: NaviKnee
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-A01677-34
Record Dates: First submitted 2021-12-14; First posted 2022-06-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single-blind, randomised, prospective comparative study in two parallel groups (conventional or computer-assisted arthroplasty).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-assisted arthroplasty (Experimental)
  Interventions: Device: Computer-assisted arthroplasty
- Conventional arthroplasty (No Intervention)

INTERVENTIONS:
Device: Computer-assisted arthroplasty — Computer-assisted arthroplasty
  Arms: Computer-assisted arthroplasty

SUMMARY:
Evaluation of a new navigation system in computer-assisted total knee arthroplasty.

DETAILED DESCRIPTION:
Single-blind, randomised, prospective comparative study in two parallel groups (conventional or computer-assisted arthroplasty).

The patient will be evaluated during 3 visits: inclusion D0 (before arthroplasty), M3 (intermediate visit 3 months after arthroplasty) and M12 (final visit 12 months after arthroplasty).

ELIGIBILITY:
Inclusion Criteria:

* Adult man or woman who has signed the informed consent for participation in the study,
* Patient with primary uni or bilateral gonarthrosis
* For whom an indication for total knee arthroplasty has been given

Exclusion Criteria:

* History of fracture, arthroplasty or osteotomy of the knee
* Severe preoperative laxity warranting a constrained prosthesis
* Inflammatory rheumatic disease or any other progressive concomitant condition that may impact on the patient's functional prognosis
* Traumatic articular or extra-articular deformities of the lower limb
* Neurological disease, after-effects of a stroke
* Mental deficiency or any other reason that may hinder the understanding or the strict application of the protocol
* Patient not affiliated to the French social security system
* Patient under legal protection, guardianship or curatorship
* Patient already included in another therapeutic study protocol or having participated in another trial in the previous three months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
KSS M12 | Month 12
  Assessment of functional outcome at 12 months by Knee Scoring System (KSS) score

SECONDARY OUTCOMES:
KSS M3 | Month 3
  Assessment of functional outcome at 3 months by Knee Scoring System (KSS) score
KOOS JR M3 | Month 3
  Functional self-evaluation of the knee joint: Knee injury and Osteoarthritis Outcome Score (KOOS)
KOOS JR M12 | Month 12
  Functional self-evaluation of the knee joint: Knee injury and Osteoarthritis Outcome Score (KOOS)
EQ-5D M3 | Month 3
  Quality of life evaluation on EuroQol 5D
EQ-5D M12 | Month 12
  Quality of life evaluation on EuroQol 5D
FJS M3 | Month 3
  Self-evaluation of patient satisfaction with Forgotten Joint Score (FJS)
FJS M312 | Month 12
  Self-evaluation of patient satisfaction with Forgotten Joint Score (FJS)
Surgery duration | Day 0
  Surgery duration
Hospitalization duration | Month 1
  Hospitalization duration
Lower limb alignment | Month 12
  Measurement of lower limb alignment in degrees of varus or valgus at M3 and M12
Postoperative outcome predictive factor | Month 1
  Description of a possible correlation between preoperative laxity and postoperative outcome
Safety analysis | Month 12
  Descriptive analysis of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Jean Mermoz, Lyon, France

IPD SHARING:
Plan to Share IPD: No